CLINICAL TRIAL: NCT03240679
Title: A Randomized Study of Biologic Scaffolds And Esophageal Healing Following Endoscopic Resection
Brief Title: Endoscopic Mucosal Resection and Cellular Matrix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty obtaining investigational product and study support.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kenneth K. Wang, Pricipal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-006909
Record Dates: First submitted 2017-04-05; First posted 2017-08-07 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Barretts Esophagus With High Grade Dysplasia; Barrett Adenocarcinoma
Keywords: Barrett's esophagus; Endoscopic Mucosal Resection
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Intervention Model Description: Pilot study 10 in each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Endoscopic submucosal resection with Extracelluar Matrix (Active Comparator): Subjects with lesions that lift and are amenable to cap-assisted endoscopic submucosal resection (EMR) will receive extracellular matrix (ECM) to the defect site.
  Interventions: Device: Acell MatriStem® Surgical Matrix
- Endoscopic submucosal resection standard of care (No Intervention): Subjects with lesions that lift and are amenable to cap-assisted endoscopic submucosal resection (EMR) will receive standard of care.

INTERVENTIONS:
Device: Acell MatriStem® Surgical Matrix — Extracellular matrix (ECM) product that is composed of collagen and natural proteins that provide a re-absorbable scaffold for tissue remodeling to facilitate constructive healing following endoscopic submucosal resection (EMR). Covers the defect site following mucosal resection using endoscopy clips or X-tac. The device will remain attached to the esophagus and integrate with native tissue over time.
  Arms: Endoscopic submucosal resection with Extracelluar Matrix

SUMMARY:
This study is being done to test the usefulness of extracellular matrix (ECM) a thin sheet placed over the site after endoscopic mucosal resection to promote healing of the esophagus.

ELIGIBILITY:
Inclusion Criteria

* Able to provide consent
* Scheduled for standard of care endoscopy that may require initial EMR evaluation of esophageal lesions
* Histological evidence of intestinal metaplasia with dysplasia or intramucosal carcinoma

Exclusion Criteria

* Pregnant women
* Prior esophageal EMR or ESD in the same region
* Anyone unable to provide informed consent
* Medical co-morbidities precluding EGD evaluation
* History of chemoradiotherapy to the neck/esophagus
* Unable to stop anticoagulation therapy (non-steroid anti-inflammatory medications are permissible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Wang, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endoscopic Submucosal Resection With Extracelluar Matrix | Endoscopic Submucosal Resection Standard of Care
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endoscopic Submucosal Resection With Extracelluar Matrix | Endoscopic Submucosal Resection Standard of Care | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Completeness of EMR Site Healing at Follow up Endoscopy
Description: Number of subjects to have complete endoscopic submucosal resection (EMR) site healing determined by the ability of the resection site to lift with saline injection during follow-up endoscopy.
Time Frame: approximately 3-4 months post EMR
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Submucosal Resection With Extracelluar Matrix | Endoscopic Submucosal Resection Standard of Care
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

2. Secondary Outcome: Presence of Stricture Formation at Follow up Endoscopy
Description: Number of subjects to have symptomatic esophageal stricture formation requiring dilation, preventing dysphagia as determined by questionnaires, and mitigating formation of post-resection scarring as determined by blinded comparison of pre- and post-resection images (taken using white-light endoscopy and electron chromoendoscopy).
Time Frame: approximately 3-4 months post EMR
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Submucosal Resection With Extracelluar Matrix | Endoscopic Submucosal Resection Standard of Care
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 16 weeks on all participants.
Arm/Group | Endoscopic Submucosal Resection With Extracelluar Matrix | Endoscopic Submucosal Resection Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Study terminated due to difficulty of obtaining investigational product and study support. Only 3 subjects accrued into the study who underwent initial endoscopy with treatment and follow-up endoscopies approximately 3 months later.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT03240679/Prot_SAP_000.pdf